CLINICAL TRIAL: NCT00353873
Title: A Multicentre, Randomised, Double-blind, Double Dummy, Parallel Group Study to Compare the Salmeterol/Fluticasone Propionate Combination (SeretideTM) at a Dose of 50/100µg Twice Daily and Fluticasone Propionate (FlixotideTM) at a Dose of 200µg Twice Daily, Both Delivered Via a Dry Powder Inhaler (DiskusTM) for 12 Weeks in Asthma in Children Aged 4-11 Years Not Controlled by Inhaled Corticosteroids Alone at Medium Dose
Brief Title: Seretide Versus Flixotide In Asthmatic Children Not Controlled By Inhaled Corticosteroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM104926
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: FLIXOTIDE; asthmatics children 4-11 years; SERETIDE; asthma-control
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone propionate (FLIXOTIDE™) (Active Comparator): Fluticasone propionate (FLIXOTIDE™) at a dose of 200μg twice daily
  Interventions: Drug: Fluticasone propionate
- Fluticasone propionate/salmeterol (SERETIDE™) (Experimental): Salmeterol/fluticasone propionate combination (SERETIDE™) at a dose of 50/100μg twice daily
  Interventions: Drug: Fluticasone propionate/salmeterol

INTERVENTIONS:
Drug: Fluticasone propionate — 200μg twice daily
  Arms: Fluticasone propionate (FLIXOTIDE™)
Drug: Fluticasone propionate/salmeterol — 50/100μg twice daily
  Other Names: Fluticasone propionate
  Arms: Fluticasone propionate/salmeterol (SERETIDE™)

SUMMARY:
This study will compare two treatment strategies (doubling the dose of inhaled steroids or adding a long acting beta2 agonist to the inhaled steroid at the same dose) in children not controlled by inhaled steroid alone at medium dose. The fixed combination SERETIDE 100/50 one inhalation twice daily will be compared to FLIXOTIDE 100 two inhalations twice daily.

DETAILED DESCRIPTION:
A multicentre, randomised, double-blind, double dummy, parallel group study to compare the salmeterol/fluticasone propionate combination (SERETIDE™) at a dose of 50/100mcg twice daily and fluticasone propionate (FLIXOTIDE™) at a dose of 200mcg twice daily, both delivered via a dry powder inhaler (DISKUS™) for 12 weeks in asthma in children aged 4-11 years not controlled by inhaled corticosteroids alone at medium dose

ELIGIBILITY:
Inclusion criteria:

* A documented clinical history of asthma for a period of at least 6 months.
* A documented history (within 12 months of Visit 1) of airway reversibility of = 15% based either on Forced expiratory volume (FEV1) or PEF measured pre and post inhalation of 200 mcg salbutamol. (If no documented history of reversibility exists, patients must demonstrate a =15% reversibility at Visit 1).
* Receiving an inhaled corticosteroid at a medium dose (beclomethasone dipropionate HydroFluoroAlkane (HFA) non fine particle = 400-500 mcg/day or beclomethasone HFA fine particle = 200mcg/day, or budesonide =400 mcg/day or fluticasone = 200 mcg/day (or fluticasone 250mcg/day if subject is taking a 125mcg MDI rather than the 100mcg Diskus), for at least 3 months prior to Visit 1 and at a stable dose for at least 4 weeks prior to Visit 1.
* Able to use the Mini-Wright peak flow meter and subject or parent/guardian had to be able to record the subject's maximum PEF correctly.
* Able to perform FEV1 correctly.
* Subject's guardian/parent able to complete an eDRC on behalf of the subject. The eDRC should be completed by the guardian/parent.
* Able to use a DISKUS™ correctly.
* At least one parent(s)/guardian(s) has to give written informed consent to participate in the study.

At the end of the run-in period (Visit 2), subjects must still meet the criteria for entry into the run-in period and also have:

* not achieved the criteria for the 'Well-controlled' asthma during two or more of the 4 weeks prior to Visit 2.

Exclusion criteria:

* Female subjects who have reached menarche.
* Received any investigational study medication in the 4 weeks prior to Visit 1.
* Experienced a respiratory tract infection in the 4 weeks prior to Visit 1.
* Experienced an acute asthma exacerbation requiring emergency room treatment within 4 weeks or hospitalisation within 12 weeks of Visit 1.
* Any use of oral/parenteral or depot corticosteroid within 12 weeks of Visit 1.
* Any use of long-acting inhaled beta2-agonists or oral beta2-agonists within 4 weeks of Visit 1.
* Any use of leukotriene antagonists or theophyllines within 4 weeks of Visit 1.
* Any known clinical or laboratory evidence of a serious uncontrolled disease (including serious psychological disorders) which is, in the opinion of the investigator, likely to interfere with the study.
* Subjects with a known or suspected hypersensitivity to inhaled corticosteroids, beta2-agonists, or any components of the formulations (e.g. lactose)
* A relative of any of the site staff, including the investigator or study co-coordinator.
* Has previously been entered into this study.

Subjects will be excluded from participating in the treatment period of the study if the following occurred during the run-in period:

* Pre-bronchodilator FEV1 <60% (assuming that measurement was correctly performed).
* Any change in asthma medication (excluding use of prophylactic study specific salbutamol for prevention of asthma symptoms due to exercise).
* Respiratory tract infection or asthma exacerbation.
* Use of oral, parenteral or depot corticosteroids.
* Emergency visit due to asthma.
* Non-compliance with the completion of the eDRC (i.e. during the 4 week period between visits, non compliance is defined as less than 5 days of completed data within any one week for four weeks - subjects must complete at least 5 days a week for the entire run-in period).

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 506 (Actual)
Dates: Start 2005-11-18 (Actual); Primary Completion 2006-10-26 (Actual); Study Completion 2006-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (58):
- Belgium (5):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Denmark (2):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Odense
- France (11):
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Grasse
  - GSK Investigational Site, Laon
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Oyonnax
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Michel
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Vaux En Velin
  - GSK Investigational Site, Villejuif
- Italy (4):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Perugia, Umbria
- Latvia (2):
  - GSK Investigational Site, Daugavpils
  - GSK Investigational Site, Riga
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Tauragė
  - GSK Investigational Site, Vilnius
- Netherlands (10):
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Beek en Donk
  - GSK Investigational Site, Deurne
  - GSK Investigational Site, Emmen
  - GSK Investigational Site, Ermelo
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Spijkenisse
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tiel
  - GSK Investigational Site, Woerden
- Norway (3):
  - GSK Investigational Site, Drammen
  - GSK Investigational Site, Kongsvinger
  - GSK Investigational Site, Oslo
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
- Russia (7):
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novokuznetsk
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Syktyvkar
  - GSK Investigational Site, Tomsk
- Spain (5):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Seville
- Sweden (2):
  - GSK Investigational Site, Sollentuna
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: SAM104926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAM104926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SAM104926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SAM104926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SAM104926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAM104926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SAM104926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 46 sites in 12 countries: Belgium (4), Denmark (1), France (8), Italy (3), Latvia (3), Lithuania (3), the Netherlands (6), Norway (1), Poland (4), Russian Federation (9), Spain (3) and Sweden (1) from 18 November 2005 to 26 October 2006.
Pre-assignment Details: A total of 584 participants were screened and entered into a 4-week run-in period receiving fluticasone propionate (FP) 100 microgram (mcg) dry powder inhaler (DISKUS) twice-daily (BD) and inhaled salbutamol as required. The number of participants randomized was 321 and 303 participants received investigational product post randomization.
Groups:
- FP 200 mcg BD: Participants received one inhalation from dry powder inhaler A (FP 100 mcg) and dry powder inhaler B (FP 100 mcg) BD, in the morning and evening for 12 weeks. Participants were provided salbutamol 100 mcg per actuation metered dose inhaler (MDI) to be used as needed throughout the study, for prevention of exercise induced asthma and symptomatic relief from asthma symptoms.
- Salmeterol/Fluticasone Propionate (SFC) 50/100 mcg BD: Participants received one inhalation from dry powder inhaler A (SFC 50/100 mcg) and dry powder inhaler B (placebo for FP 100 mcg) BD, in the morning and evening for 12 weeks. Participants were provided salbutamol 100 mcg per actuation MDI to be used as needed throughout the study, for prevention of exercise induced asthma and symptomatic relief from asthma symptoms.
Period: Overall Study
Arm/Group | FP 200 mcg BD | Salmeterol/Fluticasone Propionate (SFC) 50/100 mcg BD
Started | 153 | 150
Completed | 147 | 147
Not Completed | 6 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Exacerbation | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- FP 200 mcg BD: Participants received one inhalation from dry powder inhaler A (FP 100 mcg) and dry powder inhaler B (FP 100 mcg) BD, in the morning and evening for 12 weeks. Participants were provided salbutamol 100 mcg per actuation MDI to be used as needed throughout the study, for prevention of exercise induced asthma and symptomatic relief from asthma symptoms.
- SFC 50/100 mcg BD: Participants received one inhalation from dry powder inhaler A (SFC 50/100 mcg) and dry powder inhaler B (placebo for FP 100 mcg) BD, in the morning and evening for 12 weeks. Participants were provided salbutamol 100 mcg per actuation MDI to be used as needed throughout the study, for prevention of exercise induced asthma and symptomatic relief from asthma symptoms.
- Total: Total of all reporting groups
Arm/Group | FP 200 mcg BD | SFC 50/100 mcg BD | Total
Number analyzed (Participants) | 153 | 150 | 303
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.0 (2.01) | 8.1 (2.00) | 8.0 (2.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 53 | 108
  Male | 98 | 97 | 195
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3 | 2 | 5
  White - Arabic/North African Heritage | 4 | 4 | 8
  White - White/Caucasian/European Heritage | 146 | 144 | 290

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Morning Peak Expiratory Flow (PEF) Over 12 Weeks in Intent-to-treat (ITT) Population
Description: PEF is the maximum flow generated during expiration, as measured with a peak flow meter and recorded in electronic diary record card (eDRC), performed with maximal force and started after a full inspiration. The mean morning PEF measurement was constructed by calculating a simple mean for each participant over the interval Weeks 1 to 12. All PEF measurements were converted to the Wright/McKerow peak flow meter scale for the purposes of analyses. The change from Baseline is then calculated by subtracting the Baseline PEF values from the individual on-treatment values. Baseline was calculated as the mean of the values recorded on the seven days preceding randomization. The analysis was done using analysis of covariance (ANCOVA) adjusted for baseline PEF, country amalgamation, age, sex and treatment.
Time Frame: Baseline; Week 1 up to Week 12
Population: ITT Population: All participants randomized to treatment who received at least one dose of randomized study medication. Only participants with analyzable data at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters/Minute (L/min)
Arm/Group | FP 200 mcg BD | SFC 50/100 mcg BD
Number analyzed (Participants) | 152 | 150
Liters/Minute (L/min) | 19.3 (2.12) | 26.9 (2.13)
Statistical Analysis 1: Comparison: FP 200 mcg BD vs SFC 50/100 mcg BD; Test type: Non-Inferiority or Equivalence — Non-inferiority was tested using a one-sided significance level of 2.5%. If the lower confidence interval for the difference SFC-FP falls above -12 L/min the once daily SFC treatment combination was deemed to be statistically non-inferior. In the event that the lower confidence limit (2.5% 1-sided significance) exceeded 0, and using a separate closed testing procedure, superiority could be established; p = 0.012, ANCOVA; Mean Difference (Net) = 7.6, 95% CI 2-sided [1.7 to 13.5], Standard Error of Mean 3.01

2. Primary Outcome: Mean Change From Baseline in Morning PEF Over 12 Weeks in Per Protocol (PP) Population
Description: PEF is the maximum flow generated during expiration, as measured with a peak flow meter and recorded in eDRC, performed with maximal force and started after a full inspiration. The mean morning PEF measurement was constructed by calculating a simple mean for each participant over the interval Weeks 1 to 12. All PEF measurements were converted to the Wright/McKerow peak flow meter scale for the purposes of analyses. The change from Baseline is then calculated by subtracting the Baseline PEF values from the individual on-treatment values. Baseline was calculated as the mean of the values recorded on the seven days preceding randomization. The analysis was done using ANCOVA adjusted for baseline PEF, country amalgamation, age, sex and treatment.
Time Frame: Baseline; Week 1 up to Week 12
Population: PP Population: All participants in the ITT Population who did not have any protocol violations which could impact treatment effect. Only participants with analyzable data at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | FP 200 mcg BD | SFC 50/100 mcg BD
Number analyzed (Participants) | 135 | 127
L/min | 18.4 (2.14) | 27.7 (2.21)
Statistical Analysis 1: Comparison: FP 200 mcg BD vs SFC 50/100 mcg BD; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.003, ANCOVA; Mean Difference (Net) = 9.3, 95% CI 2-sided [3.2 to 15.3], Standard Error of Mean 3.08

3. Secondary Outcome: Number of Participants Who Achieved 'Totally Controlled' (TC) Asthma
Description: TC asthma is defined as no daily symptoms, no night-time wakening due to asthma, no exacerbations, no rescue salbutamol/albuterol use, no emergency visits, >=80% predicted morning PEF, and no treatment related adverse events enforcing a change in asthma therapy over 7 consecutive days. Number of participants/group who achieved the status of at least TC during the last 8 weeks (wks) of treatment was analyzed using logistic regression, including covariates for sex, age, treatment group, country amalgamation and baseline pre-bronchodilator Forced Expiratory Volume in one second (FEV1). Asthma control was assessed each week for the last 8 wks of treatment period. Each week was classified as 'TC', 'Well Controlled' (WC), 'Not Controlled' or 'Unevaluable'. A participant was considered to have TC asthma if they achieved 4/4, 5/5, 6/6, 6/7, 7/8 or 8/8 wks that were TC. 'Unevaluable' classification included participants with less than 4 wks of data during the assessment period.
Time Frame: Week 5 up to Week 12
Population: ITT Population. Only participants with analyzable data at the indicated time point were assessed.
Measure: Number; unit: Participants
Arm/Group | FP 200 mcg BD | SFC 50/100 mcg BD
Number analyzed (Participants) | 152 | 150
Participants | 23 | 28
Statistical Analysis 1: Comparison: FP 200 mcg BD vs SFC 50/100 mcg BD; Test type: Superiority or Other; p = 0.389, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.7 to 2.4]

4. Secondary Outcome: Number of Participants Who Achieved WC Asthma
Description: WC asthma is defined as two or more of symptom score >1 only allowed on <=2 days/week, rescue salbutamol/albuterol use on <=2 days/week and up to a maximum of 4 times per week, >=80% predicted morning PEF daily assessed for 7 consecutive days and all the following criteria: no night-time awakening due to asthma, no exacerbations, no emergency visits, no treatment related adverse events enforcing a change in any asthma therapy. Number of participants/group who achieved the status of at least WC during the last 8 wks of treatment was analyzed using logistic regression, including covariates for sex, age, treatment group, country amalgamation and baseline prebronchodilator FEV1. Each week was classified as 'WC', 'Not Controlled' or 'Unevaluable'. A participant was considered to have WC asthma if they achieved 4/4, 5/5, 6/6, 6/7, 7/8 or 8/8 wks that were WC. 'Unevaluable' classification included participants with less than 4 wks of data during the assessment period.
Time Frame: Week 5 up to Week 12
Population: ITT Population. Only participants with analyzable data at the indicated time point were assessed.
Measure: Number; unit: Participants
Arm/Group | FP 200 mcg BD | SFC 50/100 mcg BD
Number analyzed (Participants) | 152 | 150
Participants | 61 | 65
Statistical Analysis 1: Comparison: FP 200 mcg BD vs SFC 50/100 mcg BD; Test type: Superiority or Other; p = 0.535, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.7 to 1.9]

ADVERSE EVENTS:
Time Frame: Serious adverse events and non-serious adverse events were collected from the first day of treatment until the last day of treatment (up to 12 weeks).
Description: On-treatment serious adverse events and non-serious adverse events were reported for ITT Population.
Arm/Group | FP 200 mcg BD | SFC 50/100 mcg BD
Serious Adverse Events (participants affected / at risk) | 3/153 | 3/150
Other Adverse Events (participants affected / at risk) | 61/153 | 55/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FP 200 mcg BD (N=153) | SFC 50/100 mcg BD (N=150)
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Laryngotracheitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FP 200 mcg BD (N=153) | SFC 50/100 mcg BD (N=150)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Headache (Nervous system disorders) | 23 | 27
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Nasopharyngitis (Infections and infestations) | 19 | 14
Rhinitis (Infections and infestations) | 10 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.